CLINICAL TRIAL: NCT03824704
Title: A Phase 2, Open-label Study to Evaluate Rucaparib in Combination With Nivolumab in Patients With Selected Solid Tumors (ARIES)
Brief Title: A Study to Evaluate Rucaparib in Combination With Nivolumab in Patients With Selected Solid Tumors (ARIES)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor made a business decision to discontinue the study due to low accrual.
Sponsor: pharmaand GmbH (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Foundation Medicine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-338-097
Record Dates: First submitted 2019-01-21; First posted 2019-01-31 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma; High Grade Serous Carcinoma; Endometrioid Adenocarcinoma
Keywords: PARP; PARPi; PARP inhibitor; ARIES; Opdivo; Rucaparib; Nivolumab; PD-1; BRCA; LOH; CO-338; Immunotherapy; BMS-936558; Clovis; Clovis Oncology; Rubraca
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Carcinoma, Endometrioid | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A: Ovarian Cancer Cohort (Experimental): Oral rucaparib and Intravenous (IV) nivolumab (combination therapy)
  * Cohort A1
  * Cohort A2
  Interventions: Drug: Rucaparib; Drug: Nivolumab

INTERVENTIONS:
Drug: Rucaparib — Oral rucaparib will be administered twice daily
  Other Names: Rubraca; CO-338
Drug: Nivolumab — IV nivolumab will be administered once every 4 weeks
  Other Names: Opdivo; BMS-936558

SUMMARY:
This is an open label Phase 2, 2-stage, 2-cohort study to evaluate rucaparib in combination with nivolumab in patients with high-grade serous or endometroid ovarian cancer.

Patients entering the following cohorts must have BRCA mutational status confirmed by a central lab:

* Cohort A1: No BRCA mutation in tumor; high level of LOH (loss of heterozygosity)
* Cohort A2: BRCA mutation in tumor

ELIGIBILITY:
General Inclusion Criteria:

* ≥ 18 years of age
* Adequate organ function
* Life expectancy ≥ 16 weeks
* Women of childbearing potential must have a negative serum pregnancy test
* High-grade serous or endometrioid epithelial ovarian, fallopian tube, or primary peritoneal cancer
* Received 1 or 2 prior regimens, including ≥ 1 prior platinum-based therapy and have platinum-sensitive disease
* Relapsed/progressive disease (confirmed by radiologic assessment)
* Willing and able to have a biopsy of tumor at screening and after 4 weeks of treatment.
* Measurable disease (RECIST v1.1)- Cohort A1 only
* ECOG performance status of 0 to 1

General Exclusion Criteria

* Active second malignancy
* Central nervous system brain metastases
* Evidence of interstitial lung disease, active pneumonitis, myocarditis, or history of myocarditis.
* Active, known or suspected autoimmune disease (eg, autoimmune hepatitis).
* Condition requiring systemic treatment with either corticosteroids
* Prior treatment with a PARP inhibitor or immune checkpoint inhibitor.
* Non-epithelial tumors (pure sarcomas) or ovarian tumors with low malignant potential (ie, borderline tumors) or mucinous tumors. Mixed Mullerian tumors/carcinosarcomas are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen N Moore, MD, Principal Investigator — Lead Investigator for Ovarian Cohort A
Locations (5):
- United States (5):
  - Community Cancer Institute, Clovis, California
  - Memorial Health University Medical Center, Savannah, Georgia
  - Women's Cancer Care, Covington, Louisiana
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Vermont Medical Center, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 subject was recruited from 1 site in the United States. The Sponsor then discontinued the study due to low accrual.
Groups:
- Cohort A: Ovarian Cancer Cohort: Patients received combination therapy, including oral rucaparib 600mg administered twice daily starting on Cycle 1 Day 1 and intravenous (IV) nivolumab 480mg administered on Day 1 of every 4-week cycle, starting on Cycle 2 Day 1.
Period: Overall Study
Arm/Group | Cohort A: Ovarian Cancer Cohort
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by RECIST v1.1 as Assessed by the Investigator
Description: Objective response rate (ORR) is defined as the percentage of patients with a best confirmed response of complete response (CR) or partial response (PR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as assessed by the investigator.
Time Frame: From enrollment until disease progression (up to approximately 2 years)
Population: This study was discontinued by the sponsor so no data is available for this outcome measure.
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 0

2. Primary Outcome: The Effect of Rucaparib on the Immune Microenvironment
Description: Change in expression of the immune marker PD-L1 pre and post-rucaparib treatment; Cohort A2 only
Time Frame: From enrollment to primary completion of study (up to approximately 2 years)
Population: This study was discontinued by the sponsor so no data is available for this outcome measure.
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: ORR by RECIST v1.1 and Gynecological Cancer InterGroup (GCIG) Cancer Antigen 125 (CA-125 Criteria)
Description: Objective Response Rate (ORR) is defined as the percentage of patients with a best confirmed response of complete response (CR) or partial response (PR) by RECIST v1.1 as assessed by the investigator or a confirmed response per Gynecological Cancer InterGroup (GCIG) cancer antigen 125 (CA-125 criteria)
Time Frame: For patients with measurable disease, every 8 weeks after the start of combination treatment for 3 years, then every 24 weeks thereafter until disease progression or up to 25 months. Study data collection expected to last for 2 years.
Population: This study was discontinued by the sponsor so no data is available for this outcome measure.
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-Free Survival (PFS) is calculated as 1+ the number of days from the first dose of study drug to disease progression by RECIST, as determined by the investigator or death due to any cause, whichever occurs first.
Time Frame: From randomization until disease progression (up to approximately 2 years)
Population: This study was discontinued by the sponsor so no data is available for this outcome measure.
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) for any confirmed RECIST CR or PR measured from the date of the first response until the first date that progressive disease (PD) is documented.
Time Frame: For patients with measurable disease, every 12 weeks after the start of combination treatment for 3 years, then every 24 weeks thereafter until disease progression. Study data collection expected to last for 2 years
Population: This study was discontinued by the sponsor so no data is available for this outcome measure.
Arm/Group | Cohort A: Ovarian Cancer Cohort
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time informed consent was obtained until 28 days after last dose of study drug.
Description: If a subject experiences the same preferred term (system organ class) multiple times, then the subject will be counted only once for that preferred term (system organ class).
Arm/Group | Cohort A: Ovarian Cancer Cohort
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Ovarian Cancer Cohort (N=1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Ovarian Cancer Cohort (N=1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (4)
Dsypepsia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (5)
Chest pain (General disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Panic attack (Psychiatric disorders) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The Sponsor made a business decision to discontinue the study due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with investigators require proposed public disclosures of trial results to be submitted to Sponsor for review prior to publication. Sponsor may request deletion of confidential information or a delay in publication to address intellectual property concerns, but Sponsor may not suppress publication of the trial results indefinitely. Sponsor may request delay of a single-center publication until after the release of a multi-site publication or an agreed upon period of time.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03824704/Prot_SAP_000.pdf